CLINICAL TRIAL: NCT05874154
Title: Evaluation of Tibial Nerve Selective Neurotomy Compared to Botulinum Toxin Injections for Spastic Foot Treatment in Post-stroke Patients According to a Goal-centered Approach
Acronym: FOOTNEUROTOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0905
Record Dates: First submitted 2023-04-19; First posted 2023-05-24 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Post Stroke Seizure; Spastic Foot
Keywords: Tibial nerve selective neurotomy; botulinum toxin; spastic foot; post-stroke patient
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tibial nerve selective neurotomy (Experimental)
  Interventions: Procedure: Tibial nerve selective neurotomy
- Botulinum toxin injection (Active Comparator)
  Interventions: Drug: Botulinum toxin injection

INTERVENTIONS:
Procedure: Tibial nerve selective neurotomy — Patients in the STN group will undergo a pre-anaesthetic visit before surgery to validate the possibility of general anesthesia. The surgery will be performed at maximum 3 months after inclusion. The muscles that have been defined pre-randomization will be targeted by the surgery. The duration of the surgery is about 1 hour and 30 minutes.
  Arms: Tibial nerve selective neurotomy
Drug: Botulinum toxin injection — Patients in the BoNT group will be treated with BoNT A under electromyography, electrical stimulation and/or ultrasound guidance (V0). In the absence of scientific evidence between the efficacy of onabotulinumtoxin A and abobotulinumtoxin A, physician will be free to choose between these two BoNT formulation which are both authorized for the treatment of lower limb spasticity. The physician will determine the muscles targeted by the BoNT (gastrocnemius and soleus for equinus, posterior tibialis for varus, and long flexor digitorum and flexor hallucis for claw toes), the appropriate dose and dilution based on his experience, following a semi-guided table of equivalence for respective doses of onabotulinumtoxin A and abobotulinumtoxin A. A delay superior to 3 months will be respected after the last injection and the muscles that have been defined pre-randomization will be targeted by injections.
  Arms: Botulinum toxin injection

SUMMARY:
In France, more than 110.000 patients are hospitalized for stroke per year. It is the leading cause of sudden disabilities in adults. Incidence of spastic foot is evaluated at 1 year post stroke from 18% to 56% of hemiplegic patients. Spasticity, defined as an increase in the velocity-dependent response to muscle stretch measured at rest, is part of the upper motor neuron syndrome and is characterized by an increase in tonic stretch reflex. It has been proposed that upper motor neuro syndrome may induce not only spasticity but also other types of muscles overactivity such as spastic dystonia, co-contraction and clonus. In hemiplegic patients, lower limb spasticity within the posterior part of the leg frequently results in equino-varus foot and toes claw. These abnormal postures in hemiplegics may affect activities of daily living such as shoes fitting, balance, ambulation-walking, comfort (pain) and may become irreducible (tendon shortening) if not treated.

The purpose of this study is to compare the interest of each treatment (BoNT-A versus STN) in order to specify both techniques indications and up-date current guidelines of lower-limb spasticity for hemiplegic patients.

This study aims to confirm a greater reduction of calf muscles spasticity after STN as compared to BoNT-A, as observed in the only published monocentric randomized controlled trial. Our study originality is to perform a multi-center RCT with a pre-established sample size. This study will also quantify progress towards personal goals using the goal attainment scaling (GAS) and will assess other components related to the consequences of carve muscle spasticity on balance, ambulation, self-care and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (older than 18 years)
* Man and woman
* Hemiparesis secondary to stroke (delay from stroke > 1 year)
* Foot with equinovarus with or without toe claw due to spasticity of at least the triceps surae and /or one of the following muscles: tibialis posterior, flexor digitorum and hallucis longus muscles.
* Spasticity confirmed with no isolated tendon shortening diagnosed using tibialis nerve block under local anesthesia with at least a 5 degrees gain in passive or active ankle dorsal flexion.
* Covered by National French insurance
* Able to understand French and the purpose of the study
* Informed consent signed by the patient or consent obtained from a relative or trusted person of the patient

Exclusion Criteria:

* Known sensitivity to BoNT or botulinum toxin A excipients
* Contraindication to surgery under general anesthesia
* History of myasthenia
* Pregnant woman (confirmed by urinary test) or breastfeeding
* Patient under legal protection
* Patients unable to follow the requirement of the study according to the investigator or supported by a family member

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Evolution of the value of Goal Attainment Scaling | through study completion, 14 months
  Primary endpoint will be assessed using the Goal Attainment Scaling before treatment and the evaluation at the endpoint. Goals are defined before initiation of treatment, and attainment at study end is scored using a 5-point scale (-2, -1, 0, 1, 2); -2: pretreatment level, -1: less than expected; 0: expected goal; +1: somewhat more than expected; +2: best possible outcome expected

SECONDARY OUTCOMES:
Evolution of Functional outcomes | through study completion, 14 months
  Functional outcomes before treatment, at 5 weeks using Goal Attainment Scaling primary outcome scoring
Tardieu's scale | through study completion, 14 months
  Tardieu's scale assesses spasticity with movement velocity, muscle reaction angle and quality.
Modified Ashworth scale | through study completion, 14 months
  -Modified Ashworth scale, measures spasticity level according to a level scale (0,1,1+,2,3,4), 0=absence of muscle tone increase and 4=rigidity in flexion or extension of affected part(s)
Evolution of ankle motion range | through study completion, 14 months
  Active and/or passive ankle motion range Improvement at 5 weeks and endpoint
Proportion of patients with antispastic drug | through study completion, 14 months
measure of pain level | through study completion, 14 months
  Pain type using a self-rating scale for estimating the likelihood of neuropathic painscale before treatment (named DN4), at 5 weeks and endpoint using a 0 to 10 visual analogic scale
Proportion of patients with adverse event | through study completion, 14 months
  Adverse effects by systematic assessment at 5 weeks and endpoint.
Psychometric qualities of the Consumer satisfaction questionnaire (named CSQ-8) | through study completion, 14 months
  Patient reported Experience Measures will be assessed at endpoint with the CSQ-8 questionnaire
10 meter walk test - speed | through study completion, 14 months
  Walking speed with the 10 meter walk test (10MWT)
10 meter walk test - distance | through study completion, 14 months
  distance improvement assessed using the 6 minutes walking test (6MWT)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Pierre Wertheimer, Bron
  - AP-HP, Clichy
  - CHU de Nantes, Nantes
  - Hôpital Henry Gabrielle, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: No